CLINICAL TRIAL: NCT07289308
Title: The Effect of Combined Versus Sequential Attentional Focus Instructions on Upper Extremity Function in Subacute Stroke Patients: An Assessor-Blinded Randomized Controlled Trial
Brief Title: Effects of Combined vs. Sequential Attentional Focus Instructions on Upper Extremity Function in Subacute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EKPP25ST
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Upper Extremity Dysfunction; Cue, Threat
Keywords: Wolf Motor Function Test; Motor Learning; Functional Recovery; Fugl-Meyer Assessment; Action Research Arm Test
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This is a prospective, assessor-blinded, randomized controlled parallel-group study. Subacute stroke patients will be randomly assigned to one of three groups: Combined Focus of Attention Group (CFAG), Sequential Focus of Attention Group (SFAG), or Control Group (CG). Each participant will receive a standardized rehabilitation program, with the experimental groups additionally receiving task-specific upper extremity training with group-specific attentional focus instructions. Outcomes will be assessed at baseline and after four weeks by a blinded physiotherapist to evaluate the effects of combined versus sequential attentional focus instructions on upper extremity motor function.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation to ensure unbiased measurement of upper extremity function. Interventionists delivering the rehabilitation sessions are not blinded due to the need to provide group-specific attentional focus instructions. Participants are aware of the type of instructions they receive, but they are not informed of the study hypothesis or comparative group details. This single-assessor blinded design minimizes bias while maintaining intervention fidelity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Focus of Attention Group (CFAG) (Experimental): Participants in the Combined Focus of Attention Group will receive a standardized rehabilitation program plus a task-specific upper extremity training session with combined internal and external attentional focus instructions. During each task (e.g., reaching, grasping, holding objects), participants will be instructed to focus simultaneously on body movements (internal focus, e.g., "feel your shoulder moving as you extend your arm") and movement effects on the environment (external focus, e.g., "focus on the target and guide your hand to touch it"). Sessions are conducted five times per week in the clinic and twice per week at home, each lasting 60 minutes (45 minutes standard rehab + 15 minutes attentional focus training), over four weeks.
  Interventions: Other: Combined Focus of Attention Instructions; Other: standart rehabilitation program
- Sequential Focus of Attention Group (SFAG) (Experimental): Participants in the Sequential Focus of Attention Group will receive a standardized rehabilitation program plus a task-specific upper extremity training session with sequential attentional focus instructions. Internal focus cues (e.g., "feel your shoulder moving as you extend your arm") are provided during the first two weeks to enhance basic motor control, followed by external focus cues (e.g., "focus on the target and guide your hand to touch it") during the next two weeks to improve movement efficiency and functional performance. Sessions are conducted five times per week in the clinic and twice per week at home, each lasting 60 minutes (45 minutes standard rehab + 15 minutes attentional focus training), over four weeks.
  Interventions: Other: Sequential Focus of Attention Instructions; Other: standart rehabilitation program
- Control Group (Active Comparator): Participants in the Control Group will receive the standardized rehabilitation program only, without any specific attentional focus instructions. The program includes task-oriented upper extremity exercises targeting range of motion, motor control, coordination, and functional performance. Sessions are conducted five times per week in the clinic and twice per week at home, each lasting 60 minutes, over four weeks.
  Interventions: Other: standart rehabilitation program

INTERVENTIONS:
Other: Combined Focus of Attention Instructions — Participants perform task-specific upper extremity exercises while receiving simultaneous internal and external attentional focus cues, directing attention both to body movements (internal focus) and movement effects on the environment (external focus). This combined approach aims to enhance motor control, movement efficiency, and functional performance.
  Arms: Combined Focus of Attention Group (CFAG)
Other: Sequential Focus of Attention Instructions — Participants perform task-specific upper extremity exercises with internal attentional focus cues during the first two weeks (focusing on body movements, e.g., "feel your shoulder moving"), followed by external attentional focus cues during the next two weeks (focusing on movement effects, e.g., "focus on the target and guide your hand to touch it").
  Arms: Sequential Focus of Attention Group (SFAG)
Other: standart rehabilitation program — All participants receive a standardized, evidence-based rehabilitation program targeting upper extremity range of motion, motor control, coordination, and functional performance. Sessions are conducted five times per week in the clinic and twice per week at home, each lasting 45 minutes, over four weeks.

SUMMARY:
Stroke is a leading cause of long-term disability, and upper extremity impairments-affecting about 80% of survivors-limit functional reach, grasp, and manipulation more severely than lower limb deficits. Despite partial recovery of walking ability, meaningful functional use of the paretic arm remains limited. Conventional rehabilitation often lacks sufficient intensity, task specificity, and motor learning principles, highlighting the need for more effective approaches.

The subacute phase of stroke (up to 6 months post-onset) represents a period of heightened neuroplasticity and strong rehabilitation potential. During this time, integrating cognitive and motor training-such as attentional focus strategies-has gained attention. External focus enhances movement efficiency through motor automaticity, whereas internal focus supports early motor control. Evidence suggests that combining these strategies may optimize recovery, yet their relative effectiveness in stroke rehabilitation remains unclear.

Two main instructional approaches exist: combined attentional focus (internal and external cues delivered within the same session) and sequential attentional focus (internal focus first, followed by external focus as control improves). While both show therapeutic promise, comparative data in stroke populations are lacking.

This study aims to compare combined versus sequential attentional focus instructions in improving upper extremity function in subacute stroke. We hypothesize that a combined approach-starting with internal focus early, then integrating external focus-will yield superior motor improvements.

DETAILED DESCRIPTION:
Stroke is a major global cause of long-term disability. Upper extremity deficits are particularly common, affecting nearly 80% of individuals after stroke and manifesting as weakness, impaired selective motor control, abnormal muscle tone, sensory disturbances, and reduced coordination. These deficits cause substantial limitations in functional reach, grasp, and object manipulation, and they persist more severely compared with lower extremity impairments. Although most stroke survivors regain some degree of independent ambulation, only a minority recover meaningful functional use of the paretic upper limb, resulting in a disproportionately higher disability burden for the upper extremity.

Conventional rehabilitation often shows limited effectiveness in improving upper extremity outcomes because training intensity is typically insufficient, task specificity is restricted, and interventions do not consistently apply established motor learning principles. These challenges underscore the need for new therapeutic perspectives that more effectively harness neuroplasticity through high-intensity, task-oriented, and motor learning-based approaches tailored to the complex demands of upper extremity recovery.

Upper-extremity motor functions, which are often severely impaired in the acute phase of stroke, gradually begin to recover during the transition into the subacute period as spontaneous neurobiological repair processes become more active. Subacute stroke refers to the recovery phase that begins after the first week post-onset and extends through the early months, during which spontaneous biological recovery and neuroplasticity remain highly active. Although many frameworks define the core subacute window as the first 3 months, functional recovery and rehabilitation responsiveness continue meaningfully up to 6 months, which is widely accepted as the upper limit of the subacute period in clinical research and guideline-based stroke classification. Therefore, including patients within the first 6 months post-stroke ensures enrolment during a period of high rehabilitative potential.

In recent years, the integration of physical exercise and cognitive training has emerged as a promising strategy for enhancing both cognitive and motor functions in rehabilitation. One example of combining motor tasks with cognitive components is attentional focus training, which includes external and internal attentional focus strategies. External attentional focus directs the learner's attention to the effects of movement (e.g., "focus on the movement of the ball") and has been consistently shown to enhance movement efficiency and task performance. This effect is believed to occur through increased motor automaticity and reduced conscious interference. Conversely, internal attentional focus emphasizes the mechanical components of body movements (e.g.,'focus on your hand position') and can support the development of foundational motor control, particularly during the early stages of motor learning and recovery.

Recent evidence suggests that both internal and external attentional focus strategies can complement each other in therapeutic contexts. Internal focus (IF) supports early stroke rehabilitation by enhancing basic motor control, whereas external focus (EF) improves movement efficiency and functional parameters in later stages. EF has also been reported to outperform IF in improving upper extremity performance in stroke populations. These findings suggest that combining IF and EF-either simultaneously or in a structured progression-may better align with the evolving demands of stroke recovery.

In terms of enhancing upper extremity function and overall motor recovery, two primary approaches have been explored: sequential and combined attentional focus training. Combined attentional focus instruction involves delivering internal and external focus cues within the same training session or task-either concurrently or in close temporal proximity-allowing patients to benefit from both improved motor control and enhanced movement efficiency. In contrast, Sequential attentional focus instruction involves providing internal and external focus cues in a structured order-typically beginning with internal focus to establish basic motor control, followed by external focus as movement efficiency and automaticity improve. Although both approaches show promise, their comparative effectiveness has not been directly examined in stroke populations, indicating a clear need for research evaluating these instructional strategies within stroke rehabilitation.

Our primary aim is to compare the effects of combined and sequential attentional focus instructions on upper extremity motor function in patients with subacute stroke. We hypothesize that implementing combined attentional focus instructions (internal attentional focus instructions in the early stages of recovery, followed by a combination with external attentional focus instructions in later stages) will lead to greater improvements in upper extremity function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years at enrollment (Kwakkel et al., 1996; Coupar et al., 2012).
2. Stroke diagnosed by a neurologist between 1 week and 6 months before enrollment (Langhorne et al., 2020; Bernhardt et al., 2017).
3. Medically stable, as confirmed by a neurologist, with controlled and non-fluctuating vital signs (Stinear et al., 2020; Powers et al., 2019; Winstein et al., 2016).
4. Sufficient cognitive function to follow instructions, sustain attention, and actively participate in rehabilitation, as judged by the treating therapist (Stinear et al., 2020; Boyd et al., 2018).
5. Brunnstrom stage 2-5 in the affected upper limb (Brunnstrom, 1970; Langhorne et al., 2020).
6. Individuals with a Modified Ashworth Scale (MAS) score <3: Participants were required to have a MAS score of less than 3 in both the upper and lower extremities to ensure that spasticity remained at a manageable level and to allow safe participation in upper-limb motor rehabilitation (Pandyan et al., 2005; Li & Francisco, 2015; Ada et al., 2020).
7. Preserved corticospinal tract integrity, confirmed by a positive Motor Evoked Potential (MEP) response (Stinear et al., 2017; Byblow et al., 2015; Stinear et al., 2020).
8. Moderate to severe upper-extremity motor impairment, determined by Fugl-Meyer Assessment (FMA) scores of 0-47 (0-19 severe, 20-47 moderate) (Fugl-Meyer et al., 1975).

Exclusion Criteria:

* Spasticity level: Individuals with a Modified Ashworth Scale (MAS) score ≥3 in either the upper or lower extremities were excluded, as marked hypertonicity and severe spastic contractions could negatively affect proximal stabilization and movement strategies, thereby interfering with upper-limb task performance (Pandyan et al., 2005).
* Fractures: Participants with a current or recent fracture on the affected side of the body were excluded from the study.
* Botulinum toxin injections: Individuals who had received Botulinum Toxin (Botox) injections within the previous three months were excluded due to the potential effects of the intervention on muscle tone and motor performance.
* Communication disorders: Participants with motor or global aphasia, or other communication impairments that could interfere with understanding instructions or performing the required tasks, were excluded.
* Concurrent rehabilitation: Individuals who were concurrently receiving rehabilitation treatment at another facility were excluded to prevent potential confounding effects from parallel interventions (Winstein et al., 2016).
* Non-adherence to treatment sessions: Participants who failed to attend all required treatment sessions were excluded to ensure consistency and fidelity of the intervention protocol (Winstein et al., 2016).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment- Upper Extremity Subscore | baseline, four weeks after the baseline
  The Fugl-Meyer Assessment for the Upper Extremity (FMA-UE) is a validated scale used to evaluate motor control, coordination, and functional performance of the affected arm in stroke patients. Scores range from 0 to 66, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment-Total Score | baseline, four weeks after the baseline
  The Fugl-Meyer Assessment (FMA) is a validated scale widely used in stroke rehabilitation to evaluate upper extremity motor function, coordination, balance, and range of motion. Scores range from 0 to 66 for the upper extremity, with higher scores indicating better function; it allows classification of motor impairment as mild, moderate, or severe.
Action Research Arm Test | baseline, four weeks after the baseline
  The Action Research Arm Test (ARAT) is a validated scale used to assess upper limb function, including grasp, grip, pinch, and gross movements. Scores range from 0 to 57, with higher scores indicating better function, helping identify specific deficits and guide rehabilitation planning.
Wolf Motor Function Test | baseline, four weeks after the baseline
  The Wolf Motor Function Test (WMFT) is a validated tool used to assess upper extremity motor function in stroke patients, evaluating both movement quality and task completion time across functional and strength-based activities. Scores range from 0 to 75, with higher scores indicating better motor performance.

CONTACTS AND LOCATIONS:
Overall Officials: Emirhan Kocer, PT, Principal Investigator — Bahcesehir University, Graduate Education Institute; Pelin Pisirici, PT, PhD, Study Chair — Bahcesehir University, Faculty of Health Sciences
Locations (1):
- Neur-On Clinic, İstinye University, Bahcesehir Liv Hospital Stroke Center, Istanbul, Turkey (Türkiye)